CLINICAL TRIAL: NCT03776357
Title: A Rehabilitation Tool to Determine Patient's Stay in Hospital After Joint Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding halted
Sponsor: Derek Amanatullah (Other)
Responsible Party: Sponsor-Investigator, Derek Amanatullah, Assistant professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 46061
Record Dates: First submitted 2018-12-10; First posted 2018-12-14 (Actual); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Total Joint Replacement Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): The application used is build upon the company's category-defining, FDA- cleared Virtual Exercise Rehabilitation Assistant (VERA™) and create a platform that streamlines the performance and management of post-acute care physical therapy. The rehab tool will provide us with functional outcome score.
  Interventions: Device: VERA clinic

INTERVENTIONS:
Device: VERA clinic — A software system used with the Microsoft Kinect intended to support the physical rehabilitation of adults in the clinic and at home.

SUMMARY:
This is the research study of a rehabilitation tool that informs, guides and empowers clinicians to care for their patients. We hope to learn ways to improve patient outcomes, reduce costs and increase value to the healthcare system

DETAILED DESCRIPTION:
The investigator hope to learn co-relation between the rehab tool and clinical findings and analyse association if any. Rehab tool will optimize care according to the patient's specific needs and provided insights to patients length of stay in the hospital. these data driven insights will be used to observe correlation between machine and clinic data

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for Primary unilateral total joint replacement
* Patient age should be more than or equal to 18 years.
* Patient must speak English

Exclusion Criteria:

* Patients undergoing bilateral primary knee replacement surgery
* Patients undergoing revision knee replacement surgery
* No uncorrectable deformity
* No deformity greater than 15 degree
* No hip arthritis
* No wheelchair dependency
* Patients not willing and capable to sign the written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford outpatient center, Redwood City, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Participants utilize FDA cleared Virtual Exercise Rehabilitation Assistant (VERA™) platform during pre-operative visit to obtain functional outcome scores.
Period: Overall Study
Arm/Group | Experimental
Started | 9
Completed | 6
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Participants utilize the VERA platform during pre-operative visit to obtain functional outcome scores.
Arm/Group | Experimental
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Gait aide use [Count of Participants; unit: Participants] — The gait aide use ranges in the order of decreasing performance as Nothing > Cane > crutch > walker.
  Participants
    Nothing | 9
    Cane | 0
    crutch | 0
    walker | 0
Range of motion ( maximum degrees) [Mean (Standard Deviation); unit: degrees]
  Extension | 0.6 (1.7)
  Flexion | 117.8 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay in Hospital Through Discharge
Time Frame: Up to 2 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Experimental
Number analyzed (Participants) | 9
days | 2 [2 to 2]

2. Secondary Outcome: Number of Participants Requiring Gait Aid Use
Description: The gait aide use ranges in the order of decreasing performance as Nothing > Cane > crutch > walker.
Time Frame: 3 months post operative visit
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 9
Participants
  None ( no gait aide) | 9
  Cane | 0
  Crutch | 0
  Walker | 0

3. Secondary Outcome: Knee Society Score (KSS)
Description: To assess the effectiveness of the device by calculating knee society score (KSS) after surgery. The scale ranges from 0-100 with grading as Score 80-100 - Excellent Score 70-79 - Good Score 60-69 - Fair Score below 60 - Poor
Time Frame: 3 months post operative visit
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 9
Participants
  Excellent (80-100) | 6
  Good (70-79) | 0
  Fair (60-69) | 2
  Poor ( below 60) | 1

4. Secondary Outcome: Knee Range of Motion
Description: To assess the effectiveness of the device by calculating range of motion (maximum degrees)
Time Frame: 3 months post operative visit
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Experimental
Number analyzed (Participants) | 9
degrees
  extension | 1.1 (2.2)
  flexion | 107.8 (17.5)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
The study terminated early and did not meet its planned enrollment size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT03776357/Prot_000.pdf